CLINICAL TRIAL: NCT06820502
Title: OUTCOMES of SIMULTANEOUS TRANSURETHRAL PROSTATE and BLADDER TUMOR RESECTION VERSUS TRANSURETHRAL BLADDER TUMOR RESECTION in BLADDER TUMOR with BLADDER PROSTATE HYPERPLASIA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Allama Iqbal Medical College (Other)
Responsible Party: Principal Investigator, TOOBA HAMID, Post Graduate Resident, Allama Iqbal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERB179/8/23-12-2024/S1ERB
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Bladder Cancer Recurrence; BPH (Benign Prostatic Hyperplasia); Bladder Cancer
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder Neoplasms | interventions — Transurethral Resection of Prostate; Transurethral Resection of Bladder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients undergoing TURBT and TURP simultaneously (Experimental): Patients undergoing TURBT and TURP simultaneously for Bladder tumour and Benign Prostatic Hyperplexia
  Interventions: Procedure: Transurethral Resection of Prostate (TURP); Procedure: Transurethral Resection Of Bladder Tumor
- Patients undergoing TURBT (Experimental): Patients undergoing TURBT only for Bladder Tumour and BPH
  Interventions: Procedure: Transurethral Resection Of Bladder Tumor

INTERVENTIONS:
Procedure: Transurethral Resection of Prostate (TURP) — TURP:
  Transurethral resection of the prostate remains the criterion standard therapy for obstructive prostatic hypertrophy and is both the surgical treatment of choice and the standard of care when medication fails. It improves obstructive voiding symptoms and urinary flow rate with success rates ranging from 85 to 90% .
  Arms: Patients undergoing TURBT and TURP simultaneously
Procedure: Transurethral Resection Of Bladder Tumor — TURBT:
  Trans-urethral resection of bladder tumor (TURBT), performed endoscopically, is the firstline procedure for diagnosis, staging, and treatment of visible bladder tumors,

SUMMARY:
The rationale of my study is that studies have shown that between 50% and 70% of patients treated with trans-urethral bladder tumor resection (TURBT) alone for NMIBC have recurrence with stage and grade progression in 10% to 15% and because of this theoretical danger of tumor cell implantation, many urologists avoid simultaneous trans-urethral prostate resection (TURP) and TURBT due to fear of implantation of tumor cells in the denuded areas of the resected prostate and prefer to perform a separate procedure for each pathological condition. However, others observed no deleterious effects of simultaneous TURBT and TURP. This unsettled controversy that has spanned almost 4 decades. This study will delineate guidelines for outcome of these procedures in terms of better prognosis for patients.

OBJECTIVE:

The objective of the study is to compare the outcome of simultaneous trans-urethral bladder tumor and prostate resection versus trans-urethral bladder tumor resection alone in bladder tumor with prostate hyperplasia in terms of in terms of recurrence of bladder tumor SUBJECTS AND METHODS Study Design: Randomized controlled trial Settings: Department of Urology, Jinnah Hospital and Allama Iqbal Medical College, Lahore.

Study Population: Patients who will undergo TURP and TURBT at Jinnah Hospital, Lahore will be study population.

Duration of study: 3 months after approval of synopsis. Sampling Technique: Non-Probability / consecutive Sampling Sample Size: Sample size calculated with 80 % power of study and 5 % level of significance Assumed recurrence rate of simultaneous trans-urethral bladder tumor resection with prostate resection (Group A) = 53.6% Assumed recurrence rate of trans-urethral bladder tumor resection alone (Group B) = 86.9% Required sample size of total of 60 patients (30 patients in each group)

SAMPLE SELECTION:

Inclusion Criteria

* Males aged 40 - 65 year
* First diagnosis of bladder neoplasm less than 4 cm, confined in urinary bladder
* Prostate volume ≥ 40 and ≤ 80 ml with normal PSA level and obstructive voiding symptoms Exclusion Criteria

  * Patients with previous prostatic, urethral surgery and urinary bladder surgery like diverticulectomy, ureteric reimplant in urinary bladder
  * Patients with coagulopathy
  * Previous history of heart diseases
  * Diagnosis of prostate cancer
  * Urethral stenosis, previous pelvic irradiation, and neurogenic bladder.
  * Recurrent Bladder Tumor

DATA COLLECTION PROCEDURE:

The study involves 60 male patients diagnosed with bladder carcinoma, meeting inclusion criteria. Informed consent, emphasizing data confidentiality, will be obtained. Patients will be thoroughly examined at Jinnah Hospital Lahore. Preoperative assessment includes medical history, physical examination, digital rectal examination, PSA assay, and IPSS. Patients will be randomly assigned one of two treatments through a computer aided randomization. Patients will be followed with preoperative protocols, and undergo procedures under spinal anesthesia. In group A trans-urethral resection with a resectoscope is employed for both TURBT and TURP. In Group B TURBT, a wire loop electrode through the cystoscope removes bladder tumors in small pieces. TURP involves the resectoscope removing prostate tissue in small fragments, controlled by electrocautery. Post-surgery, complications were dealt with. Tissue fragments are sent to the lab for histopathological analysis. Follow-ups adhere to EAU guidelines, recording recurrence and UTI presence. Histopathology reports follow the 2004 WHO classification. The primary outcome recurrence rate will be noted in 3 months. All the information will be collected in a structured questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 40 - 65 year
* First diagnosis of bladder neoplasm less than 4 cm, confined in urinary bladder
* Prostate volume > 40 and < 80 ml with normal PSA level and obstructive voiding symptoms

Exclusion Criteria:

-Patients with previous prostatic, urethral surgery and urinary bladder surgery Iike diverticulectomy, ureteric reimplant in urinary bladder Patients with coagulopathy Previous history of heart diseases Diagnosis of prostate cancer Urethral stenosis, previous pelvic irradiation, and neurogenic bladder. Recurrent Bladder Tumor

Ages: 40 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate is the organ in the male genital system specifically, its absent in females
Enrollment: 60 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Bladder Tumor Recurrence | after 3 months of surgery
  RECURRENCE OF TUMOUR:
  Recurrence refers to the return of bladder cancer after initial treatment. It can occur in the remaining bladder tissue (if partial cystectomy was performed), in the area where the bladder was removed or in nearby lymph nodes. Recurrence will be measured through regular follow-up cystoscopies and imaging studies (such as ct scans) as recommended by EAU guidelines. Any suspicious findings will be biopsied and confirmed through histopathology. It will be assessed after three months of surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology and Renal Transplant, Jinnah Hospital Lahore/ Allama Iqbal Medical College, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes